CLINICAL TRIAL: NCT02776982
Title: Influence of Central Obesity on the Esophageal Epithelial Barrier
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prasad G. Iyer, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-001069
Record Dates: First submitted 2016-05-16; First posted 2016-05-19 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Gastroesophageal Reflux; GERD
Keywords: Gastroesophageal reflux disease; GERD; Barrett's Esophagus; Esophageal adenocarcinoma
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research procedures (Other): Participants enrolled in study will have confocal endomicroscopy, research biopsies, mucosal impedance, and Bravo ambulatory pH capsule performed at the time of clinically indicated endoscopy.
  Interventions: Procedure: Confocal endomicroscopy; Procedure: Mucosal impedance; Procedure: Research biopsies; Procedure: Bravo ambulatory pH monitor

INTERVENTIONS:
Procedure: Confocal endomicroscopy — Confocal endomicroscopy will be performed during clinically indicated endoscopy.
Procedure: Mucosal impedance — Mucosal impedance will be performed at the time of clinically indicated endoscopy.
Procedure: Research biopsies — Research biopsies will be obtained during clinically indicated endoscopy.
Procedure: Bravo ambulatory pH monitor — Bravo ambulatory pH capsule will be placed during clinically indicated endoscopy.

SUMMARY:
This study is being done to help understand why some people with an increased amount of central obesity, without gastroesophageal reflux, develop changes to the lining of their esophagus that can potentially lead to esophageal adenocarcinoma (cancer).

ELIGIBILITY:
Inclusion Criteria:

Participants who are undergoing clinically indicated upper endoscopy with Bravo ambulatory pH capsule (off reflux medications for 7 days), in the Esophageal Clinic at Mayo Clinic.

Exclusion Criteria:

1. Pre-existing or suspected Barrett's Esophagus (> 1cm of columnar mucosa in esophagus on endoscopy
2. Oral anticoagulation precluding endoscopic biopsies
3. Patients with known hypersensitivity to fluorescein sodium.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Compare intercellular space dilation as a marker for apical junction complex integrity in esophageal squamous epithelium by using transmission electron microscopy in those patients with/without gastroesophageal reflux and with/without central obesity. | One year

SECONDARY OUTCOMES:
Compare paracellular permeability of esophageal squamous epithelium by measuring mucosal impedance and IV fluorescein leak using a confocal laser endomicroscope in those patients with/without gastroesophageal reflux and with/without central obesity. | One year
Compare the prostaglandin E2 level as measured by enzyme immunoassay in esophageal squamous epithelium in those patients with/without gastroesophageal reflux and with/without central obesity. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G Iyer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gibbens YY, Lansing R, Johnson ML, Blevins CH, Katzka DA, Iyer PG. Effects of Central Obesity on Esophageal Epithelial Barrier Function. Am J Gastroenterol. 2021 Jul 1;116(7):1537-1541. doi: 10.14309/ajg.0000000000001196. PMID 33955725
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials